CLINICAL TRIAL: NCT00575991
Title: Effect of CLA Supplementation on Body Fat Accretion Among Children Who Are Overweight or at Risk of Overweight
Brief Title: Effect of Conjugated Linoleic Acid on Body Fat in Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Bunge Loders Croklaan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H2006-0300
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Overweight
Keywords: conjugated linoleic acid, body fat, children, overweight
MeSH Terms: conditions — Overweight | interventions — Linoleic Acids, Conjugated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Dietary Supplement: Conjugated linoleic acid
- B (Placebo Comparator)
  Interventions: Dietary Supplement: Conjugated linoleic acid

INTERVENTIONS:
Dietary Supplement: Conjugated linoleic acid — 3 grams per day of 80% CLA in safflower oil (2.4 grams active CLA isomers in triglyceride form)

SUMMARY:
The prevalence of overweight children has increased dramatically over the last decade, and many overweight children will remain overweight as adults. Conjugated linoleic acid (CLA), a naturally occurring dietary fatty acid, has shown promising results in reducing body fat among adults, and we propose to test the efficacy of CLA supplementation on body fat accretion in 6 to 10 year old children who are overweight or at risk of overweight.

ELIGIBILITY:
Inclusion Criteria:

* age 6 to 10 years
* body mass index greater than 85th percentile
* Tanner stage I

Exclusion Criteria:

* medical condition
* dairy allergy

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
body composition using DXA | 6 months

SECONDARY OUTCOMES:
blood chemistry variables including fasting glucose and insulin, lipids, and liver enzymes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dale A Schoeller, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Department of Nutritional Sciences, Madison, Wisconsin, United States